CLINICAL TRIAL: NCT01184092
Title: Phase 1, Open-Label, Randomized, Single-Dose, 3-Treatment, 3-Period, Cross-Over, Bioequivalence Study Comparing Phase 2b, Phase 3 And Commercial Image Tablet Formulations Of Tasocitinib (CP-690,550) Under Fasted Conditions
Brief Title: A Study To Compare The Amount Of Tasocitinib (CP-690,550) That Is Absorbed Into The Blood Of Healthy Subjects Following Oral Administration Of Three Different Tablet Versions Of Tasocitinib (CP-690,550)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A3921075
Record Dates: First submitted 2010-08-16; First posted 2010-08-18 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Bioequivalence; healthy volunteer study; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Sequence 1 (Experimental)
  Interventions: Drug: Treatment A; Drug: Treatment B; Drug: Treatment C
- Sequence 2 (Experimental)
  Interventions: Drug: Treatment A; Drug: Treatment C; Drug: Treatment B
- Sequence 3 (Experimental)
  Interventions: Drug: Treatment B; Drug: Treatment C; Drug: Treatment A
- Sequence 4 (Experimental)
  Interventions: Drug: Treatment B; Drug: Treatment A; Drug: Treatment C
- Sequence 5 (Experimental)
  Interventions: Drug: Treatment C; Drug: Treatment A; Drug: Treatment B
- Sequence 6 (Experimental)
  Interventions: Drug: Treatment C; Drug: Treatment B; Drug: Treatment A

INTERVENTIONS:
Drug: Treatment A — Single oral dose of 10 mg tasocitinib citrate (CP-690,550-10)administered as one 10 mg immediate release tablet (ICH -commercial image tablet).
  Arms: Sequence 1
Drug: Treatment B — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg immediate release filmcoated tablets (Phase 3 tablets).
  Arms: Sequence 1
Drug: Treatment C — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg tablets (Phase 2B tablets).
  Arms: Sequence 1
Drug: Treatment A — Single oral dose of 10 mg tasocitinib citrate (CP-690,550-10)administered as one 10 mg immediate release tablet (ICH -commercial image tablet).
  Arms: Sequence 2
Drug: Treatment C — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg tablets (Phase 2B tablets).
  Arms: Sequence 2
Drug: Treatment B — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg immediate release filmcoated tablets (Phase 3 tablets).
  Arms: Sequence 2
Drug: Treatment B — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg immediate release filmcoated tablets (Phase 3 tablets).
  Arms: Sequence 3
Drug: Treatment C — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg tablets (Phase 2B tablets).
  Arms: Sequence 3
Drug: Treatment A — Single oral dose of 10 mg tasocitinib citrate (CP-690,550-10)administered as one 10 mg immediate release tablet (ICH -commercial image tablet).
  Arms: Sequence 3
Drug: Treatment B — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg immediate release filmcoated tablets (Phase 3 tablets).
  Arms: Sequence 4
Drug: Treatment A — Single oral dose of 10 mg tasocitinib citrate (CP-690,550-10)administered as one 10 mg immediate release tablet (ICH -commercial image tablet).
  Arms: Sequence 4
Drug: Treatment C — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg tablets (Phase 2B tablets).
  Arms: Sequence 4
Drug: Treatment C — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg tablets (Phase 2B tablets).
  Arms: Sequence 5
Drug: Treatment A — Single oral dose of 10 mg tasocitinib citrate (CP-690,550-10)administered as one 10 mg immediate release tablet (ICH -commercial image tablet).
  Arms: Sequence 5
Drug: Treatment B — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg immediate release filmcoated tablets (Phase 3 tablets).
  Arms: Sequence 5
Drug: Treatment C — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg tablets (Phase 2B tablets).
  Arms: Sequence 6
Drug: Treatment B — Single oral dose of 10 mg CP-690,550 -10 administered as two 5 mg immediate release filmcoated tablets (Phase 3 tablets).
  Arms: Sequence 6
Drug: Treatment A — Single oral dose of 10 mg tasocitinib citrate (CP-690,550-10)administered as one 10 mg immediate release tablet (ICH -commercial image tablet).
  Arms: Sequence 6

SUMMARY:
In this study, a 10 mg dose of tasocitinib (CP-690,550) will be given to study subjects on three separate occasions using one of three different tablet formulations (tablet versions) each time. The amount of tasocitinib (CP-690,550) available in the blood following administration of each tablet formulation will be measured and compared. The overall aim of the study is to establish that a similar amount of tasocitinib (CP-690,550) is absorbed into the blood following administration of the same dose of each different tablet formulation.

DETAILED DESCRIPTION:
This is a pivotal bioequivalence study for tasocitinib (CP-690,550).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female (non-childbearing potential) subjects between the ages of 21 and 55 years, inclusive.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight for males>50 kg (110 lbs). For females, total body weight >45 kg (99 lbs).
* No evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB).

Exclusion Criteria:

* Evidence of any clinically significant illness, medical condition, or disease.
* Evidence or history of any clinically significant infections within the past 3 months.
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
PK parameters: AUCinf, AUClast and Cmax of tasocitinib (CP-690,550). | PK blood samples out to 24 hours post dose in each period

SECONDARY OUTCOMES:
PK parameters: Tmax, t½ of tasocitinib (CP-690,550). | Derived from PK blood samples out to 24 hours post dose in each period.
Safety: laboratory tests. | Pre-dose on Day 0 for Period 1 and at 24 hours post last dose in Period 3.
Safety: vital signs | Prior to dosing in each period and at 24 hours post last dose in Period 3.
Safety: adverse event reporting | Throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921075&StudyName=A%20Study%20To%20Compare%20The%20Amount%20Of%20Tasocitinib%20%28CP-690%2C550%29%20That%20Is%20Absorbed%20Into%20The%20Blood%20Of%20Healthy%20Subjects%20Following%20Oral%20Adm